CLINICAL TRIAL: NCT02066480
Title: Improved Screening for Osteoporosis in Women Between 50 and 80 Years Hospitalized in Hospital Departmental Vendee
Brief Title: Improved Screening for Osteoporosis
Acronym: ADOV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD 086-13
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women between 50 and 80 years hospitalized in CHD Vendée

SUMMARY:
Osteoporosis is a disease characterized by skeletal fragility due to decreased bone mass and deterioration of bone microarchitecture , leading to increased fracture risk for low trauma, such as spinal fractures or femoral neck .

It is estimated that 3 million people are living in France , particularly women , with an incidence that increases with age .

This disease is a major public health issue in terms of morbidity and mortality , costs and risk of recurrence (after a first fracture episode) , including risk factors are identified.

However, although bone densitometry is a reliable diagnostic tool and preventive treatments are at our disposal, screening for osteoporosis is still insufficient .

The objective of our study is to improve the detection of osteoporosis in Hospital Departmental Vendee , using a simple questionnaire seeking risk factors followed by bone densitometry or if risk factors are found. Based on the results , the patient will be sent in rheumatology consultation for implementation of treatment if necessary .

Therefore included women hospitalized in medical services , gynecology, surgery and orthopedics Hospital Departmental Vendee , aged 50 to 80 years. Will not be included women who could answer a simple questionnaire and those previously treated for osteoporosis or have already received a bone density there is less than 3 years old .

ELIGIBILITY:
Inclusion Criteria:

* Women between 50 and 80 years
* Hospitalized
* In health services, orthopedics, gynecology, surgery
* Able to respond to an easy questionnaire
* Able to give their agreement to participate in the study

Exclusion Criteria:

* Patients with dementia
* Patients can not express
* Patients at end of life
* Patients previously treated for osteoporosis or recent densitometry (BMD) <3 years
* Patients could not be seen in time by the nurse during their hospitalization
* Patients receiving a measure of legal protection

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women between 50 and 80 years hospitalized CHD Vendée
Sampling Method: Non-Probability Sample
Enrollment: 3226 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of patients screened at risk for osteoporosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire CORMIER, PH, Principal Investigator — Centre hospitalier départemental Vendée
Locations (1):
- Centre hospitalier départemental Vendée, La Roche-sur-Yon, France

REFERENCES:
- [Background] Maville M, Cormier G, Rabiller S, Dimet J, Cozic C. [Nurses mobilised in screening for osteoporosis]. Rev Infirm. 2016 Dec;65(226):42-44. doi: 10.1016/j.revinf.2016.09.016. French. PMID 27908478